CLINICAL TRIAL: NCT03848624
Title: CUHK Jockey Club HOPE 4 Care Programme - Interactive FES Cycling System
Brief Title: CUHK Jockey Club HOPE 4 Care Programme - FES Bike
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019.016
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycling Group (Experimental): Intention driven motor-assisted voluntary cycling with electrical stimulation
  Interventions: Device: Cycling Group

INTERVENTIONS:
Device: Cycling Group — Electrical pulses from a stimulator can stimulate the target muscles to generate muscle contraction to support a continuous cycling motion

SUMMARY:
The Hong Kong Jockey Club Charities Trust has supported CUHK to launch a three-year project 'CUHK Jockey Club HOPE4Care Programme' to implement four evidence-based advanced rehabilitation technologies in 40 local elderly day care centres and rehabilitation centres, to benefit the community.

Our research team had developed the "Interactive FES Cycling System" that can be used as tools for rehabilitation by individuals who have suffered from a stroke or elderly. The system can integrate both motor power and muscle power in order to facilitate an active rehabilitative exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic brain injury or intracerebral haemorrhage shown by magnetic resonance imaging or computed tomography after the onset of stroke;
* Significant gait deficit (Functional Ambulatory Category, FAC<4 [person cannot walk independently]).

Exclusion Criteria:

* Any additional medical or psychological condition that would affect their ability to comply with the study protocol, e.g., a significant orthopaedic or chronic pain condition, major post-stroke depression, epilepsy, artificial cardiac pacemaker / joint;
* Severe hip, knee or ankle contracture that would preclude passive range of motion of the leg (MAS<3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Lower-Extremity | Three months after the last training session
  Fugl-Meyer Assessment for Lower-Extremity (FMA-LE), consists of 34-level cumulative scoring system to examine lower-limb functions of hemiplegic stroke patients quantitatively through a set of lower-limb movement tasks in reflex, flexor/extensor synergy, volitional movement, coordination and speed (Fugl-Meyer, et al., 1975). All assessment items are either scoring "full", "partial", or "none" functionality in the affected side, which minimizes ceiling and floor effects. FMA-LE demonstrated high internal consistency and a reliable assessment tool for a group of 140 hemiplegic community dwelling patients (Park & Choi, 2014).

SECONDARY OUTCOMES:
6 Minute Walk Test | Three months after the last training session
  Six-Minute Walk Test (SMWT), measures the maximum walking distance covered in fixed duration as a sub-maximal test of endurance and aerobic capacity. The measurement of 6MWT is highly correlated to FAC (Mehrholz, et al., 2007) with good reliability (ICC=0.94-0.96) (Steffen, Hacker & Mollinger, 2002).
Timed 10-meter Walk Test | Three months after the last training session
  Timed 10-Meter Walk Test (10mWT), measures comfortable and fast walking speeds in short distance. The ability to increase walking speed above a comfortable pace suggests the capability to adapt to varying environments, such as crossing street, with high reliability (ICC=0.90-0.96) (Flansbjer, et al., 2005). Average walking speed of healthy elderly subjects ranges in 0.6m/s-1.4m/s, and can increase to 21%-56% above the comfortable pace for faster walking speed.
Berg Balance Scale | Three months after the last training session
  Berg Balance Scale (BBS), consists of 56-level measures to examine balance ability and to predict falling risk with high reliability (ICC=0.98) (Steffen, Hacker & Mollinger, 2002). Stroke patients were assessed based on their performance on 14 simple mobility tasks, including transfer, standing, and reaching.
Modified Ashworth Scale | Three months after the last training session
  Modified Ashworth Scale (MAS), consists of 4-level scale to examine joint spasticity based on muscle tone and resistance detected during passive stretching with good inter-rater reliability (ICC =0.85) (Bohannon & Smith, 1987).
Functional Ambulation Category Test | Three months after the last training session
  Functional Ambulatory Category (FAC) is a reliable measurement of independent walking ability on level-ground walking and stair ambulation, which is a good prediction of independent community walking post-stroke (Mehrholz, et al., 2007). FAC consists of 6-level scale: patients with FAC=4 requires supervision in level ground walking, FAC=5 requires supervision only when walking on non-level surface such as stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No